CLINICAL TRIAL: NCT05823909
Title: A Randomized, Multicenter Study of the Safety and Performance of Fabian PRICO for Saturation Targeting With Non-invasive Respiratory Support
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vyaire Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 100-P0310
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Insufficiency Syndrome of Newborn

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: fabian Therapy evolution ventilators with PRICO (Predictive Intelligent Control of Oxygenation) — 12 hours Automated PRICO FiO2 control
Device: fabian Therapy evolution ventilators with manual FiO2 control — 12 hours Manual PRICO FiO2 control

SUMMARY:
This study is planned as a part of the post market clinical follow-up (PMCF) on a CE marked product. The purpose of this study is to assess, in a routine clinical environment at two centers the use of fabian-PRICO with noninvasive ventilation and its safety and performance at targeting and maintaining accurate SpO2 levels.

DETAILED DESCRIPTION:
This is a randomized cross-over study. Subjects will be assigned to two, nominally 12-hour interventions, one with standard manual titration of FiO2 and the other with automated adjustment (PRICO). The order of these two interventions will be random.

In addition to the ventilators data, basic demographics (i.e., gestational age, birth weight, age, weight at study) of the participating infants will be recorded in the eCRF.

This study has no additional follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the neonatal unit that require non-invasive respiratory support and supplemental oxygen provided by fabian Therapy evolution ventilator
* <37 + 0 weeks gestation
* <10 kg at study entry
* FiO2 > 0.25
* Informed consent form obtained as per EC requirements

Exclusion Criteria:

* Not expected to complete 24 hours of non-invasive respiratory support
* Congenital anomalies
* Uncontrolled hemodynamics
* Severe airflow obstruction
* Intracranial hypertension
* Start of caffeine therapy within 12 hours
* Attending physician does not believe participation in the study is in the patient's best interest

Ages: 0 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Members of the Investigational team will periodically review records to identify and maintain a pool of potential investigation candidates from the NICU. It is anticipated that this pool will be significantly larger than capacity of the team to enroll into the investigation.
  The parents of potential candidates will be approached for discussion and consent prior to the desired intervention.
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Target Range Compliance | 12 hours
  Percentage of time that SpO2 is between 90-95% or above 95% when FiO2 = 21%

SECONDARY OUTCOMES:
Avoidance of SpO2 Extremes | 12 hours
  Percentage of time that SpO2 is a) <80% and b) >98% when FiO2>21%

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Ventura, MD, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori; Gianluca Lista, MD, Principal Investigator — Buzzi Children's Hospital
Locations (2):
- Italy (2):
  - Buzzi Children's Hospital, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza

IPD SHARING:
Plan to Share IPD: No